CLINICAL TRIAL: NCT05096273
Title: Retraining and Control Therapy (ReACT): Sense of Control and Catastrophic Symptom Expectations as Targets of a Cognitive Behavioral Treatment for Pediatric Psychogenic Non-epileptic Seizures (PNES)
Brief Title: Retraining and Control Therapy (ReACT): Sense of Control and Symptom Expectations as Targets of a Treatment for PNES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Fobian, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-151001004-2; R61MH127155 (NIH)
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Convulsion, Non-Epileptic
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Intervention Model Description: Children with PNES and matched controls will be prospectively enrolled.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers who conduct baseline and follow-up visits will be blinded to the condition (booster or no booster) to which the patient has been assigned. The statistician and data manger will be blinded to treatment condition when analyzing data. The PI and therapists will be blinded to participant's baseline target scores.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- CPT- Pain relief lotion (Experimental): During the initial visit participant will do the cold pressor test twice to assess catastrophic symptom expectations. After completing the 1st CPT, participants will be randomized to receive a pain relief lotion or pain sensitivity lotion. Participants will then repeat the CPT with the lotion applied to their hand.
  Interventions: Behavioral: ReACT
- CPT- Pain sensitivity lotion (Experimental): During the initial visit participant will do the cold pressor test twice to assess catastrophic symptom expectation. After completing the 1st CPT, participants will be randomized to receive a pain relief lotion or pain sensitivity lotion. Participants will then repeat the CPT with the lotion applied to their hand.
  Interventions: Behavioral: ReACT
- ReACT for PNES- Booster therapy sessions (Active Comparator): After completing the 12 therapy sessions, half of the participants will be randomized to receive 2 booster therapy sessions, 3 months and 9 months after the 12th ReACT treatment session.
  Interventions: Behavioral: ReACT
- ReACT for PNES- No Booster therapy sessions (Experimental): After completing the 12 ReACT treatment sessions, half of the participants will be randomized to not receive the 2 booster therapy sessions.
  Interventions: Behavioral: ReACT
- Healthy Control (No Intervention): Healthy controls are matched to participants with PNES based on age (+ or - 1 year), gender, race and family income. Healthy controls and their parent come for 1 baseline laboratory visit and a follow up visit 13 weeks after the baseline visit. These visits will be identical to baseline and follow-up visits of children with PNES.

INTERVENTIONS:
Behavioral: ReACT — ReACT is a novel cognitive behavioral treatment and is a PNES intervention that targets sense of control and catastrophic symptom expectations
  Other Names: Retraining and Control Therapy
  Arms: CPT- Pain relief lotion; CPT- Pain sensitivity lotion; ReACT for PNES- Booster therapy sessions; ReACT for PNES- No Booster therapy sessions

SUMMARY:
The purpose of this study is to assess sense of control and catastrophic symptom expectations as targets for Retraining and Control Therapy (ReACT- an intervention focused on changing behaviors and thoughts) for treatment of pediatric psychogenic non-epileptic seizures (PNES, episodes resembling epileptic seizures but with no medical explanation). 11-18-year-olds diagnosed with PNES will engage in twelve sessions of ReACT. Sense of control over actions will be measured by the magic and turbulence task, a well-validated measure of sense of control. Participants will complete the cold pressor test (CPT) in which participants hold their hand in cool water for as long as possible up to 3 minutes. Catastrophic symptom expectations in response to the CPT will be measured by Pain Catastrophizing Scale for Children (PCS-C) pain tolerance (time with hand in water) and cortisol response. Target assessments will occur 7 days before treatment, 7 days after 8th treatment session and 7 days after 12th treatment session. Participants will also complete long term follow-up visits via HIPAA-compliant Zoom at 6 months and 12 months after the 12th treatment session where participants will complete questionnaires. PNES frequency will be measured from 30 days before to 12 months after treatment.

DETAILED DESCRIPTION:
PNES participants and their parent come to our laboratory for a baseline visit, 2 follow-up visits and 12 therapy sessions. Participants will complete 2 long-term follow-up visits at 6 months and 12 months after the 12th treatment session via HIPAA-compliant Zoom. Half of the participants will be randomized to receive 2 booster therapy sessions after treatment. Participants must provide EEG results indicating a diagnosis of psychogenic non-epileptic seizures.

During the initial visit, participants and their parent will complete several questionnaires assessing demographics, mood and suicidality, relationships with friends and family, as well as past and current PNES symptoms. They will also complete the childhood trauma questionnaire. The treatment targets (sense of control and catastrophic symptom expectations), will be measured by the magic and turbulence computer task and pain tolerance, PCS-C and cortisol response to the CPT, respectively. After completing the CPT, participants will be randomized to receive a pain relief lotion or a pain sensitivity lotion. Participants will then repeat the CPT with the lotion applied to their hand. PNES diaries will be completed to assess PNES frequency over the previous 30 days. The baseline lab visit will last about 3 hours. Saliva will be collected over 3 time points before and after each CPT to measure cortisol response to the CPT. Participants will also collect 2 saliva samples 24 hours later to serve as a baseline outside of the laboratory setting. Participants will also be given a Respironics Actiwatch Spectrum Pro to track sleep and PNES episode severity and frequency for the 1 week between the baseline visit and first ReACT session.

All participants will then be scheduled to return in one week for their first of 12 sessions of ReACT. Before beginning the first ReACT session, participants will complete the Flanker Inhibitory Control and Attention, List Sorting Working Memory, Pattern Comparison Processing Speed, Dimensional Change Card Sort, and Picture Sequence Memory subtests. This first session will last a maximum of two hours, and the following 11 sessions will be scheduled weekly and will each last one hour. The following 11 sessions are currently conducted via telehealth due to COVID-19. Participants will be mailed another Respironics Actiwatch Spectrum Pro before the 11th therapy session to track sleep and PENS episode severity and frequency for the 2 weeks between the 11th therapy session and the lab visit one week after the 12th treatment session.

To assess treatment dose, participants will return for post lab visits one week after the 8th treatment session and 12th treatment sessions to perform tasks and fill out questionnaires completed at baseline. Long-term follow-up at 6 months and 12 months after treatment will also be conducted to assess FS frequency and questionnaires. Participants will complete the Flanker Inhibitory Control and Attention, List Sorting Working Memory, Pattern Comparison Processing Speed, Dimensional Change Card Sort, and Picture Sequence Memory subtests at the lab visit after the 12th treatment session. Each of these sessions will last about 1 to 2 hours. PNES frequency will be measured from 30 days before treatment to 12 months after treatment through PNES diaries completed by the parent and the participant.

After treatment, half of the participants will be randomized to receive 2 booster therapy sessions at 3 months and 9 months after the end of treatment. Each of these sessions will last one hour.

Healthy controls are matched to participants with PNES based on age (+ or - 1 year), gender, race and family income. Healthy controls and their parent come for a baseline laboratory visit and a follow up visit 13 weeks after the baseline visit. The baseline and follow-up appointments for healthy controls will be identical to the visits for children with PNES.

ELIGIBILITY:
Inclusion Criteria:

* 9-18 years old.
* Diagnosis of psychogenic non-epileptic seizures by a medical doctor using video-EEG.
* Family member (parent if a minor) willing to participate and that the subject with PNES chooses.

Exclusion Criteria:

* Comorbid Epilepsy
* Less than 4 PNES per month
* Other paroxysmal nonepileptic events (e.g. episodes related to hypoxic-ischemic phenomena, sleep disorders or migraine-associated disorders)
* Participation in other therapy
* Severe intellectual disability
* Severe mental illness (delusions/hallucinations)

Exclusion for CPT:

* Blood pressure >130/80 mmHg for adolescents greater than or equal to 13 years old
* Either systolic and/or diastolic blood pressure greater than or equal to 95% based on sex and age for children less than 13 years old

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Magic and turbulence task | 7 months
  Measure of perceived sense of control in response to tasks in which control is manipulated; Greater negative numbers indicate improved understanding of control. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Pain catastrophizing scale for children- situation specific | 7 months
  Measures catastrophic symptom expectations; score ranges from 0-52, higher scores indicate greater levels of pain-related anxiety. Assessment done after performing Cold Pressor Test. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Pain tolerance (time) | 7 months
  Measures catastrophic symptom expectations. Measured by the total time the participant can keep their hand in cool water during the Cold Pressor Test. Shorter time indicates less pain tolerance. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Salivary cortisol response to Cold Pressor Test | 7 months
  Measures catastrophic symptom expectations. Measured before and after the cold pressor test. Increased cortisol response indicate increased perceived pain severity. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Pain Rating Scale | 7 months
  Measures perceived pain severity after the CPT; score ranges from 0-100. Higher scores indicate greater perceived pain severity. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Stroop task | 7 months
  Measure of cognitive inhibition and selective attention, higher scores means poorer cognitive inhibition and selective attention. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).

SECONDARY OUTCOMES:
PNES Frequency | 16 months
  Measured by Psychogenic Non-epileptic Seizures (PNES) diary, including frequency, premonitory symptoms, description of PNES symptoms and duration. Assessed 30 days before treatment to 12 months after the 12th treatment session (about 16 months total).
  Frequency and severity also measured by Respironics Actiwatch Spectrum Pro. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
Pain Catastrophizing Scale for Children (PCS-C)- General | 16 months
  Measures catastrophic symptom expectations; score ranges from 0-52, higher scores indicate greater levels of pain-related anxiety. Assessment done before performing Cold Pressor Test. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Children's Somatic Symptoms Inventory (CSSI-24) | 16 months
  General somatic symptom complaints, higher scores indicate greater somatic complaints. Scores range from 0-140. Completed by participant and parent. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Anxiety Sensitivity Index (ASI) | 16 months
  Assesses catastrophic symptom expectations; higher scores indicate greater anxiety. Completed by participant and parent. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Shipley | At baseline
  Assesses verbal IQ; higher scores indicate greater verbal IQ. Completed by participant at the baseline visit.
Quality of Life in Epilepsy for Adolescents (QOLIE-AD-48) | 16 months
  Assesses health-related quality of life for children with epilepsy (used in PNES participants by instructing them to consider their PNES when asked about "seizures"); score ranges from 0-100, higher scores indicate better functioning and well-being. Completed by participant. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Sense of Agency Scale | 16 months
  Single question which asks "How much control do you believe you have over your PNES?". Completed by participant. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
LEVEL 2-Somatic Symptom report adapted from the Participant Health Questionnaire Physical Symptoms | 16 months
  Measures symptom severity in children; higher scores indicate greater symptom severity. Completed by participant and parent. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Functional Disability Inventory (FDI) | 16 months
  Completed by child and parent to measure physical functioning and disability in children with chronic pain; score ranges from 0-60, higher scores indicate greater perceived functional disability. Completed by participant and parent. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
The Impact on Family Scale | 16 months
  Assesses parental perceptions of the impact of a child's medical condition on the family; higher scores indicate greater financial burden on the family. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Childhood Trauma Questionnaire | At Baseline
  History of physical, sexual and/or emotional abuse and physical and emotional neglect, higher scores indicate greater abuse/neglect. Completed by participant at baseline visit.
The Revised Children's Anxiety and Depression Scale (RCADS) | 16 months
  Measures anxiety and depression symptoms in children; higher scores indicate increased symptom severity. Completed by participant and parent. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
The Columbia Suicide Severity Rating Scale (C-SSRS) | 16 months
  Measure that addresses the full range of suicidal thoughts and behaviors that suggest a person is at heightened risk of committing suicide. Completed by trained research study coordinator. Assessed at baseline visit, 1 week after the 8th therapy session, 1 week, 6 months and 12 months after the final therapy sessions (about 16 months total).
Healthcare Related Stigma Questionnaire | At Baseline
  Measures stigma in patients and their parents related to their interaction with health care providers; higher scores indicate greater stigma. Completed by participant and parent. Assessed at baseline visit.
COVID-19 Functional Neurological Disorders (FND) Questionnaire | At Baseline
  Assesses the effect of COVID-19 diagnosis in FND patients. Completed by Children. Assessed at baseline visit
Flanker Inhibitory Control and Attention Subtest | 4 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures executive function and attention; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session and 1 week after 12th therapy session (about 4 months total).
List Sorting Working Memory Subtest | 4 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures working memory; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session and 1 week after 12th therapy session (about 4 months total).
Pattern Comparison Processing Speed Subtest | 4 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures processing speed; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session and 1 week after 12th therapy session (about 4 months total).
Dimensional Change Card Sort Subtest | 4 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures executive function; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session and 1 week after 12th therapy session (about 4 months total).
Picture Sequence Memory Subtest | 4 months
  Subtest of the National Institute of Health Toolbox Cognition Battery. Measures episodic memory; higher scores indicate better performance. Completed by children. Assessed at 1st therapy session and 1 week after 12th therapy session (about 4 months total).
Sleep Duration | 4 months
  Measures total sleep duration in a 24-hour day. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
Sleep Efficiency | 4 months
  Measures quality of sleep. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
Sleep Onset Latency | 4 months
  Refers to the time it took the child to fall asleep after lying down in bed. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
Sleep - Bed Time | 4 months
  Measures total time in bed in a 24-hour day. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 5 months total).
Sleep - Wake Time | 4 months
  Measures total awake time in a 24-hour day. Objectively measured using Respironics Actiwatch Spectrum Pro and subjectively measured using sleep diaries. Worn/completed by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
PNES Episode Frequency | 4 months
  Measures the total number of PNES episodes the child had in a day. Objectively measured using Respironics Actiwatch Spectrum Pro. Worn by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
PNES Episode Duration | 4 months
  Measures the duration of a PNES episode. Objectively measured using Respironics Actiwatch Spectrum Pro. Worn by children. Assessed for 1 week between baseline visit and 1st therapy session and 2 weeks between 11th therapy session and 1 week after 12th therapy session (about 4 months total).
Child Self-Report Tic Questionnaire | 16 months
  Assesses intensity and frequency of motor and vocal tics reported by children at baseline and follow-up visits.
Parent Tic Questionnaire | 16 months
  Assesses intensity and frequency of motor and vocal tics experienced by children. Parent completes this questionnaire at baseline and follow-up visits.
Yale Global Tic Severity Scale | 6 months
  Assesses intensity and frequency of motor and vocal tics experienced by children. Completed by therapist at 1st therapy session and 12th therapy session.

CONTACTS AND LOCATIONS:
Locations (1):
- Sparks Center Office of Psychiatric Research, Birmingham, Alabama, United States